CLINICAL TRIAL: NCT04183803
Title: Robotic Assistance for Tunnel Positioning in Anterior Cruciate Ligament Reconstruction
Acronym: MIRRACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0029
Record Dates: First submitted 2019-11-21; First posted 2019-12-03 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior cruciate ligament; reconstruction; robot; tunnel
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rosa robot assistance (Experimental): Patients with ACL rupture requiring surgical treatment will be included. The reconstruction will be performed with hamstring tendon graft or patellar tendon graft. The femoral and tibial tunnels placement will be guided by the Rosa robot (Zimmer®).
  Interventions: Procedure: anatomic anterior cruciate ligament (ACL) reconstruction

INTERVENTIONS:
Procedure: anatomic anterior cruciate ligament (ACL) reconstruction — The reconstruction will be performed with hamstring tendon graft or patellar tendon graft. The femoral and tibial tunnels placement will be guided by the Rosa robot (Zimmer®).

SUMMARY:
Accurate ideal graft tunnel positioning is essential for the successful application of anatomic anterior cruciate ligament (ACL) reconstruction. The accurate insertion of the tibial tunnel (TT) and femoral tunnel (FT) remain a challenge.

A robotic assisted new strategy for drill TT and FT in ACL reconstruction will be performed and its efficacy and accuracy will be assess.

The investigators will prospectively include 30 patients with ACL rupture requiring surgical treatment. The reconstruction will be performed with hamstring tendon graft or patellar tendon graft. The femoral and tibial tunnels placement will be guided by the Rosa robot (Zimmer®).

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at CHU Amiens-Picardie for ACL reconstruction by practitioner who has robot experience.
* children and adults from 10 to 45 years old

Exclusion Criteria:

* Patients managed by another ACL reconstruction technique
* Patients under guardianship, curators deprived of liberty
* Pregnant and nursing women.
* Patient who refused to participate in the study and to sign informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of tunnel positioning | Day 0; during the operation
  Accuracy of tunnel positioning will be evaluated by comparing the theoretical intraoperative position and the actual post-operative position by image fusion

SECONDARY OUTCOMES:
Range of motion of the knee | day 0, during operation
  Range of motion of the knee will be measured with IKCD score (International Knee Documentation Committee) IKCD score : The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Range of motion of the knee | up to 2 years; during follow-up
  Range of motion of the knee will be measured with IKCD score (International Knee Documentation Committee) IKCD score : The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Range of motion of the knee | up to 2 years; during follow-up
  Range of motion of the knee will be measured with Lysholm (Lysholm Knee Score)
  Lysholm Knee Score : measure the domain of functioning in sports and recreational activities. This scale consists of eight items. It is scored on a scale of 0 to 100, with higher scores indicating fewer symptoms and higher levels of functioning.
Range of motion of the knee | day 0, during operation
  Range of motion of the knee will be measured with Lysholm (Lysholm Knee Score)
  Lysholm Knee Score : measure the domain of functioning in sports and recreational activities. This scale consists of eight items. It is scored on a scale of 0 to 100, with higher scores indicating fewer symptoms and higher levels of functioning.
Range of motion of the knee | up to 2 years; during follow-up
  Range of motion of the knee will be measured with ACL-RSI (Psychological ACL-RSI Score).
  Psychological ACL-RSI Score : measure patient psychological impact. This test includes 12 questions. Higher score describes no knee pathology.
Range of motion of the knee | day 0, during operation
  Range of motion of the knee will be measured with ACL-RSI (Psychological ACL-RSI Score).
  Psychological ACL-RSI Score : measure patient psychological impact. This test includes 12 questions. Higher score describes no knee pathology.
Knee stability | day 0; during operation
  Knee stability will be measured with manual test : "pivot shift"
Knee stability | day 0; during operation
  Knee stability will be measured with manual test : radiography images.
Knee stability | up to 2 years; during follow-up
  Knee stability will be measured with manual test : "pivot shift"
Knee stability | up to 2 years; during follow-up
  Knee stability will be measured with manual test : radiography images.

CONTACTS AND LOCATIONS:
Overall Officials: François Deroussen, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No